CLINICAL TRIAL: NCT04088617
Title: The Effects of Exogenous Ketones on Glucose Tolerance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H16-01846-B
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Dietary Supplement: Ketone Supplement; Dietary Supplement: Placebo

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Placebo masked with flavouring and participants consume in opaque containers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone monoester (Experimental): Acute morning dose of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate (0.45 ml/kg body weight)
  Interventions: Dietary Supplement: Ketone monoester
- Placebo (Placebo Comparator): Acute morning dose of flavour-matched placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone monoester — Acute ingestion of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate prior a 2-hour high carbohydrate mixed meal tolerance test.
  Arms: Ketone monoester
Dietary Supplement: Placebo — Acute ingestion of a taste-matched placebo prior a 2-hour high carbohydrate mixed meal tolerance test.
  Arms: Placebo

SUMMARY:
The ketone body beta-hydroxybutyrate is produced during prolonged fasting or when endogenous carbohydrate stores are depleted and can be used as an alternative fuel source. Exogenous beta-hydroxybutyrate, in the form of a ketone monoester, is proposed to have glucose-lowering potential but this has not been adequately studied. The purpose of this study is to determine whether supplementing with an acute dose of ketone monoester can improve the glycemic response to a high carbohydrate mixed meal in young healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy individuals
* Not taking any medications affecting glucose metabolism

Exclusion Criteria:

* Competitive endurance athlete (i.e., train specifically for cycling, triathlon or distance running and compete at a high level)
* Diagnosed with the chronic medical condition that may impact consumption of carbohydrates or supplements (e.g., diabetes, heart disease)
* Are currently using medications that may interfere with insulin sensitivity
* Adhere to a strict high-fat low-carbohydrate or ketogenic diet (within the last 3 months)
* Are currently using ketone supplements
* Unable to travel to and from the university in order to make your testing appointments.
* Unable to follow the controlled diet instructions required for the study.
* If pregnant or are planning to become pregnant during the study (if female)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-01-05 (Actual)

PRIMARY OUTCOMES:
Glucose area under the curve | 2-hour
  Area under the curve for glucose during high carbohydrate mixed meal tolerance test

SECONDARY OUTCOMES:
Insulin area under the curve | 2-hour
  Insulin area under the curve during high carbohydrate mixed meal tolerance test
Free fatty acids area under the curve | 2-hour
  Non-esterified fatty acids area under the curve during high carbohydrate mixed meal tolerance test
Glucose incremental area under the curve | 2-hour
  Incremental area under the curve (above baseline) for glucose during high carbohydrate mixed meal tolerance test
Insulin incremental area under the curve | 2-hour
  Incremental area under the curve (above baseline) for insulin during high carbohydrate mixed meal tolerance test
2-hr glucose level | 2-hour
  Plasma glucose assessed 2-hr after high carbohydrate mixed meal tolerance test
Beta-hydroxybutyrate level | 2-hour
  Blood beta-hydroxybutyrate concentration assessed by handheld monitor

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No